CLINICAL TRIAL: NCT01255306
Title: The Influence of Silicone Oil on Nerve Fiber Layer Thickness After Pars Plana Vitrectomy
Status: Completed | Type: Observational
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Mia Zoric Geber, Mia Zoric Geber, MD, University Hospital Sestre Milosrdnice
Other Study IDs: KBSM-30-1/10
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Results first posted 2012-01-24 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Rhegmatogenous Retinal Detachment; Toxic Effect of Silicone; Glaucoma Due to Silicon Oil
Keywords: Rhegmatogenous retinal detachment; Pars plana vitrectomy; Silicone oil; Retinal nerve fibre layer
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NO IOP: Patients without raised IOP
  Interventions: Other: Optical coherence tomography
- RAISED IOP: Patients with raised IOP
  Interventions: Other: Optical coherence tomography; Drug: Local medical treatment of raised intraocular pressure

INTERVENTIONS:
Other: Optical coherence tomography — Optical coherence tomography will be performed in all study patients following pars plans vitrectomy and silicone oil tamponade. A fellow eye of each patient will serve as a control. Each patient enrolled in a study will receive 4 measurements:
  1. On 7th postoperative day
  2. On 30th postoperative day
  3. On 90th postoperative day
  4. On 180th postoperative day
  Other Names: Cirrus HD OCT ( Carl Zeiss Meditec, Dublin, CA )
Drug: Local medical treatment of raised intraocular pressure — In patients with raised intraocular pressure following medications will be employed in order to control the intraocular pressure:
  Cosopt (dorzolamide hydrochloride-timolol maleate ophthalmic solution; b.i.d.) Ganfort (Bimatoprost, timolol maleate ophthalmic solution; once daily) Alphagan (Brimonidine ophthalmic solution; b.i.d.) In patients with intraocular pressure less than 27 mmHg Alphagan will be prescribed. In patients with intraocular pressure greater than 27 mmHg either Cosopt, or Ganfort will be prescribed under the discretion of treating physician. If intraocular pressure in patients treated with either Cosopt or Ganfort does not drop under 21 mmHg, Alphagan will be added.
  Other Names: 1. Cosopt; 2. Ganfort; 3. Alphagan
  Groups: RAISED IOP

SUMMARY:
The aim of the study is to evaluate the influence of silicone oil on thickness of the retinal nerve fiber layer by using optical coherence tomography (OCT) in patients following pars plana vitrectomy.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the influence of silicone oil on thickness of the retinal nerve fiber layer by using optical coherence tomography (OCT) in patients following pars plana vitrectomy.

The study will include 60 patients with a temporary silicone oil tamponade who will be surgically treated with pars plana vitrectomy for rhegmatogenous retinal detachment and proliferative vitreoretinopathy. All subjects will be subdued to complete ophthalmologic examinations, measurements of the retinal nerve fiber layer thickness by an OCT examination, tests of the visual field with the use of an Octopus computed perimeter (automated static perimetry) and FDT-perimetry - both prior to the surgery, and on control visits for check-up during the postoperative period.

All results provided by postoperative examinations will be compared with one another.

The study is expected to provide data on the effect of the silicone oil on thickness of the retinal nerve fiber layer. It is also planned to show possibilities and advantages of OCT as a method of choice in the follow-up of patients with intraocular silicone oil tamponade.

ELIGIBILITY:
Inclusion Criteria:

- patients with rhegmatogenous retinal detachment

Exclusion Criteria:

* preexistent glaucoma
* previous retinal surgery
* placement of scleral buckle during surgery
* patients with more than 1/2 of emulsified silicone oil in anterior chamber postoperatively
* patients who develop silicone oil keratopathy postoperatively
* patients who develop silicone oil cataract which blocks visualization of posterior segment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary care clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mia Zoric Geber, MD, Principal Investigator — University department of Ophthalmology, University Hospital "Sestre milosrdnice"
Locations (1):
- University Department of Ophthalmology, University Hospital "Sestre milosrdnice", Vinogradska 29, Zagreb, Croatia

REFERENCES:
- [Background] Honavar SG, Goyal M, Majji AB, Sen PK, Naduvilath T, Dandona L. Glaucoma after pars plana vitrectomy and silicone oil injection for complicated retinal detachments. Ophthalmology. 1999 Jan;106(1):169-76; discussion 177. doi: 10.1016/S0161-6420(99)90017-9. PMID 9917800
- [Background] Al-Jazzaf AM, Netland PA, Charles S. Incidence and management of elevated intraocular pressure after silicone oil injection. J Glaucoma. 2005 Feb;14(1):40-6. doi: 10.1097/01.ijg.0000145811.62095.fa. PMID 15650603
- [Background] Mastropasqua L, Carpineto P, Ciancaglini M, Falconio G, Harris A. Reproducibility of nerve fiber layer thickness measurements using optical coherence tomography in silicone oil-filled eyes. Ophthalmologica. 2001 Mar-Apr;215(2):91-6. doi: 10.1159/000050836. PMID 11244337
- [Background] Leung CK, Cheung CY, Weinreb RN, Qiu Q, Liu S, Li H, Xu G, Fan N, Huang L, Pang CP, Lam DS. Retinal nerve fiber layer imaging with spectral-domain optical coherence tomography: a variability and diagnostic performance study. Ophthalmology. 2009 Jul;116(7):1257-63, 1263.e1-2. doi: 10.1016/j.ophtha.2009.04.013. Epub 2009 May 22. PMID 19464061
- [Background] Kee C, Cho C. Evaluation of retinal nerve fiber layer thickness in the area of apparently normal hemifield in glaucomatous eyes with optical coherence tomography. J Glaucoma. 2003 Jun;12(3):250-4. doi: 10.1097/00061198-200306000-00012. PMID 12782844
- [Background] Wollstein G, Schuman JS, Price LL, Aydin A, Beaton SA, Stark PC, Fujimoto JG, Ishikawa H. Optical coherence tomography (OCT) macular and peripapillary retinal nerve fiber layer measurements and automated visual fields. Am J Ophthalmol. 2004 Aug;138(2):218-25. doi: 10.1016/j.ajo.2004.03.019. PMID 15289130
- [Background] Shah NN, Bowd C, Medeiros FA, Weinreb RN, Sample PA, Hoffmann EM, Zangwill LM. Combining structural and functional testing for detection of glaucoma. Ophthalmology. 2006 Sep;113(9):1593-602. doi: 10.1016/j.ophtha.2006.06.004. PMID 16949444
- [Background] Yalvac IS, Altunsoy M, Cansever S, Satana B, Eksioglu U, Duman S. The correlation between visual field defects and focal nerve fiber layer thickness measured with optical coherence tomography in the evaluation of glaucoma. J Glaucoma. 2009 Jan;18(1):53-61. doi: 10.1097/IJG.0b013e318179f751. PMID 19142136
- [Background] Inoue M, Iriyama A, Kadonosono K, Tamaki Y, Yanagi Y. Effects of perfluorocarbon liquids and silicone oil on human retinal pigment epithelial cells and retinal ganglion cells. Retina. 2009 May;29(5):677-81. doi: 10.1097/IAE.0b013e318196fca1. PMID 19174720
- [Derived] Zoric Geber M, Bencic G, Vatavuk Z, Ivekovic R, Friberg TR. Retinal nerve fibre layer thickness measurements after successful retinal detachment repair with silicone oil endotamponade. Br J Ophthalmol. 2015 Jun;99(6):853-8. doi: 10.1136/bjophthalmol-2014-305839. Epub 2014 Dec 15. PMID 25510920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a diagnosis of retinal detachment who fulfilled enrolment criteria were included in the study. All patient were enrolled through University Department of Ophthalmology, University Hospital "Sestre milosrdnice".
  The recruitment started in April 2010 and the last patient was enrolled in June 2011.
Pre-assignment Details: We excluded one patient who developed severe inflammatory reaction 5 days following pars plana vitrectomy and silicone oile tamponade from the study.
Period: Overall Study
Arm/Group | NO IOP | RAISED IOP
Started | 26 | 33
Completed | 25 | 32
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NO IOP | RAISED IOP | Total
Number analyzed (Participants) | 26 | 33 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 25 | 36
  >=65 years | 15 | 8 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 63.80 (12.97) | 58.21 (12.26) | 60.67 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 10 | 22 | 32
Region of Enrollment [Number; unit: participants]
  Croatia | 26 | 33 | 59

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Retinal Nerve Fibre Layer Thickness Change Measured by Optical Coherence Tomography
Description: Retinal nerve fiber layer thickness change measured by optical coherence tomography might be an additional parameter that could provide new insights into clinical decision making in patients with silicone oil tamponade.
Time Frame: 6 months
Population: We included all patients that have completed necessary follow up visits and have had optical coherence tomography measurements at all visits in the final analysis.
Measure: Mean (Standard Deviation); unit: micrometer
Units Other Than Participants: eyes
Groups:
- STUDY EYES: Study eyes that underwent pars plana vitrectomy and silicone oil tamponade
- CONTROL EYES: Fellow eye of each patient
Arm/Group | STUDY EYES | CONTROL EYES
Number analyzed (Participants) | 57 | 57
Number analyzed (eyes) | 57 | 57
micrometer
  RNFL thickness at 7th postop. day | 96.23 (16.39) | 87.07 (10.79)
  RNFL thickness at 30th postop. day | 96.09 (21.59) | 87.93 (11.14)
  RNFL thickness at 90th postop. day | 97.56 (23.72) | 87.37 (11.51)
  RNFL thickness at 180th postop. day | 100.40 (23.35) | 88.93 (11.67)

2. Secondary Outcome: Retinal Nerve Fiber Layer Thickness Change in Patients With Raised Intraocular Pressure Secondary to Silicone Oil Endotamponade
Description: To assess whether retinal nerve fiber layer thickness changes in patients with raised intraocular pressure secondary to silicone oil endotamponade.
Time Frame: 6 months
Population: We included all patients who completed follow up visits and who had valid OCT measurements as defined per protocol.
Measure: Mean (Standard Deviation); unit: micrometer
Units Other Than Participants: eyes
Groups:
- CONTROL: Fellow eye of each patient
Arm/Group | NO IOP | RAISED IOP | CONTROL
Number analyzed (Participants) | 25 | 32 | 57
Number analyzed (eyes) | 50 | 64 | 57
micrometer
  RNFL thickness at 7th postop. day | 96.08 (15.18) | 96.34 (17.51) | 87.07 (10.79)
  RNFL thickness at 30th postop. day | 93.76 (17.65) | 97.91 (24.35) | 87.93 (11.14)
  RNFL thickness at 90th postop. day | 96.44 (23.08) | 98.44 (24.53) | 87.37 (11.51)
  RNFL thickness at 180th postop. day | 101.76 (23.00) | 99.34 (23.93) | 88.93 (11.67)

ADVERSE EVENTS:
Arm/Group | STUDY EYES | CONTROL EYES
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No